CLINICAL TRIAL: NCT05129345
Title: Addressing Barriers to Achieving Cardiometabolic Disorders Prevention and Treatment Goals for Persons Living With HIV in the Southeastern United States
Brief Title: Addressing Barriers to Achieving Cardiometabolic Disorders Prevention and Treatment Goals for PLWH in the SE US
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108897
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Dyslipidemias; Type 2 Diabetes; HIV-1-infection
Keywords: Hypertension; Dyslipidemias; Type 2 Diabetes; HIV-1-infection
MeSH Terms: conditions — Hypertension; Dyslipidemias; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1: People living with HIV who are at least 35 years of age and who have one or more of the following conditions: hypertension, dyslipidemia, or type 2 diabetes. All genders, races and ethnicities will be included in this study. Subjects will have a telephone visit including being consented electronically and complete a demographic survey, a photography training visit and an interview visit.
- Aim 2: People living with HIV who are at least 35 years of age and who have one or more of the following conditions: hypertension, dyslipidemia, or type 2 diabetes. All genders, races and ethnicities will be included in this study. Subjects will have a telephone visit and be electronically consented to study and complete an electronic survey.
- Aim 3: Group composed of 10 willing participants recruited from the participating clinics and community based organizations and may include, HIV providers, nurses, pharmacists, people living with HIV who have cardiometabolic disorders, and representatives of the community advisory boards, and any other key stakeholders. There will be 3 one hour meetings over 3 months.

SUMMARY:
This study has 3 aims. Aim 1: Identify social determinants of cardiometabolic health and determine facilitators and modifiable barriers in achieving treatment goals.

Aim 2: Assess PLWH knowledge, skills, and confidence for self-management of cardiometabolic disorders.

Aim 3: Tailor a self-management support and education intervention with stakeholder input to address barriers to achieving treatment goals for cardiometabolic disorders in PLWH at the study sites.

DETAILED DESCRIPTION:
Aim 1: 20 PLWH ages 35 years and older with at least one cardiometabolic disorder (hypertension, dyslipidemia, or type 2 diabetes) will participate in in-depth interviews (IDIs) using photo elicitation to capture the social environment and contextual determinants of cardiometabolic disorders for PLWH. Prior to IDIs, PLWH will take photographs of facilitators and barriers to reaching their cardiometabolic health goals. During IDIs we will discuss the content of the photographs and explore the most salient facilitators and barriers that an intervention (Aim 3) must address to achieve treatment goals for cardiometabolic disorders at the study sites.

Aim 2: 120 PLWH with the same eligibility criteria as Aim 1 across the study sites will complete a Patient Activation Measure survey to assess knowledge, skills, and confidence for self-management of their cardiometabolic disorders. Logistic regression models will assess the predictors of knowledge, skills and confidence for self management of these disorders in order to inform the tailoring of the intervention in Aim 3.

Aim 3: Guided by the Behavior Change Wheel model and using the human-centered design approach, we will engage key stakeholders (healthcare providers, community advisory board members, and PLWH with cardiometabolic disorders) in the tailoring of a self-management support and education intervention that has been found to be effective in the general population. We will engage stakeholders in an iterative process spanning three months by first developing understanding of the self-management and education intervention, reviewing the results from Aim 1 and 2 and brainstorming possible tailoring options within the context in which PLWH live and receive care in order to arrive at an intervention that is desirable, feasible, and viable. A final recommendation of the tailored intervention will be presented to the participating HIV providers, Ending the HIV Epidemic Committee in Mecklenburg County, and the Duke Center for AIDS Research Community Advisory Board. The completion of these aims will provide the data for publication, an adapted evidence-based intervention, and community and healthcare collaborations necessary to launch an R21 application to assess the acceptability, fidelity, and appropriateness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2

* People living with HIV who are at least 35 years of age and who have one or more of the following conditions: hypertension, dyslipidemia, or type 2 diabetes.

Aim 3

* Participants recruited from the participating clinics and community based organizations and may include, HIV providers, nurses, pharmacists, people living with HIV who have cardiometabolic disorders, and representatives of the community advisory boards, and any other key stakeholders. Age 18 or older.

Exclusion Criteria:

* Those who don't understand English and those who are blind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aims 1 and 2
  * People living with HIV who are at least 35 years of age and who have one or more of the following conditions: hypertension, dyslipidemia, or type 2 diabetes.
  Aim 3
  * Participants recruited from the participating clinics and community based organizations and may include, HIV providers, nurses, pharmacists, people living with HIV who have cardiometabolic disorders, and representatives of the community advisory boards, and any other key stakeholders. Age 18 or older.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Number of social determinants of cardiometabolic health identified from interviews | 2 weeks after enrollment
  Interviews with PLWH who have cardiometabolic disorders to determine salient barriers and facilitators of achieving treatment goals for cardiometabolic disorders
Aim 2: Patient engagement in healthcare as measured by the Patient Activation Measure (PAM) | Baseline
  Assess PLWH knowledge, skills, and confidence for self-management using the PAM which is a 13 item survey, Likert scale from strongly disagree to agree strongly.
Aim 3: Number of strategies modified in the self-management support and education | Up to 3 months
  Tailoring of self-management support and education intervention using stakeholder engagement strategies

CONTACTS AND LOCATIONS:
Overall Officials: Charles Muiruri, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University - Charlotte Study Sites, Charlotte, North Carolina
  - Duke University - Duke Study Site, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No